CLINICAL TRIAL: NCT05876364
Title: A Phase 1, Dose-escalation, Multi-center, Open-label, Study to Evaluate the Safety, Reactogenicity and Immunogenicity of a Preventive SARS-CoV-2 Vaccine (QTP104) in Healthy Adults
Brief Title: Study to Assess Safety, Reactogenicity and Immunogenicity of the repRNA(QTP104) Vaccine Against SARS-CoV-2(COVID-19)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Quratis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CT-QTP104-002
Record Dates: First submitted 2023-05-01; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: mRNA Vaccine; Replicon mRNA; Self-replicating mRNA
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): Injection in the muscle at 0day , 28 day
  Interventions: Biological: QTP104 1ug
- Cohort 2 (Experimental): Injection in the muscle at 0day , 28 day
  Interventions: Biological: QTP104 5ug
- Cohort 3 (Experimental): Injection in the muscle at 0day , 28 day
  Interventions: Biological: QTP104 25ug

INTERVENTIONS:
Biological: QTP104 1ug — Intramuscular injections of 1 µg of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (QTP104) on days 1 and 28
  Arms: Cohort 1
Biological: QTP104 5ug — Intramuscular injections of 5 µg of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (QTP104) on days 1 and 28
  Arms: Cohort 2
Biological: QTP104 25ug — Intramuscular injections of 25 µg of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (QTP104) on days 1 and 28
  Arms: Cohort 3

SUMMARY:
This study is to evaluate the safety, reactogenicity, and immunogenicity of the QTP104 vaccine against SARS-CoV-2 infection in healthy adults.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, immunogenicity of 3 doses of QTP104. The reason for including 3 doses were to further explore the immunogenicity of these dose levels. This clinical trial is an open label and does not apply to randomized assignment procedures. This study is an open label and does not apply to the maintenance and release procedure of double-blinding. The selection of healthy adults is to confirm the safety of dose-escalation through phase 1 clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female aged 19 to 55 years at the screening visit (Visit 1)
2. Subject with a Body Mass Index (BMI) of 18kg/m2 or more and 30kg/m2 or less at the screening visit (Visit 1)
3. Women of childbearing potential who have not undergone sterilization must agree to use an appropriate method of contraception* during this clinical trial period and up to 3 months after the end of administration of the investigational drug and there must be evidence of non-fertility at the screening visit (Visit 1)
4. Men who has not undergone a vasectomy must consent to the use of barrier contraception (i.e., condoms) and if both subejct and partner agree to use an appropriate method of contraception for the duration of the clinical trial and up to 6 months after the end of investigational drug administration
5. Subject who can collect blood and urine during this clinical trial period including the last visit
6. Subject who havs heard the detailed explanation of this clinical trial, have voluntarily decided to participate, and have agreed in writing to abide by the precautions
7. Subject who agrees not to donate blood or transfusion (including whole blood, plasma components, platelet components and platelet plasma components) during the clinical trial period

Exclusion Criteria:

[Current disease and medical history]

1. Subject who has identified any acute, chronic, or clinically significant disease as a result of a physical or laboratory examination during a screening visit (Visit 1)
2. Subject who has a history of malignant tumors within the past 5 years
3. Subject who has an immune dysfunction, including immunodeficiency disease, or a family history thereof through a medical history and/or physical examination
4. Subject who has positive SARS-CoV-2 IgG Ab results during screening visit (Visit 1)
5. Subject previously diagnosed with COVID-19
6. Subject with any acute, chronic, or clinically significant disease as a result of physical examination or laboratory examination at the screening visit (Visit 1)
7. Subject with a history of malignancy within 5 years before the first dose of the investigational drug (except for basal cell and squamous cell carcinoma of the skin)
8. Subject with immune dysfunction including immunodeficiency disease through medical history and/or physical examination, or with a family history
9. Subject with a positive result of virus test (hepatitis B test, hepatitis A test, human immunodeficiency virus test, hepatitis C test) at the screening visit (Visit 1)
10. Subject who are significantly abnormal clinically in laboratory tests, electrocardiogram, chest, and X-rays performed at the screening visit (Visit 1) and those who are judged impossible to participate in the clinical trial at the discretion of the investigator
11. Subject with a history of hypersensitivity or severe allergic reaction to vaccine administration [e.g. anaphylaxis, Guillain-Barre syndrome, urticaria*, other clinically significant reactions requiring medical intervention]
12. Urticaria: Those with a history of systemic urticaria within 5 years before administration of investigational drugs
13. Subject with diseases on such systems as hepatobiliary, kidney, nervous system (central or peripheral), respiratory (asthma, pneumonia, etc.), endocrine (uncontrolled diabetes mellitus, hyperlipidemia, etc.), cardiovascular (congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension) etc.), urinary, psychiatric, musculoskeletal disorders or have a clinically significant history that it is judged to be unable to participate in a clinical trial under the judgment of the investigator
14. Subject with autoimmune diseases including autoimmune hypothyroidism and psoriasis
15. Subject with suspected or history of alcohol or substance abuse 12 months prior to the scheduled screening visit (Visit 1). Alcohol abuse standards are defined as follows:
16. Subject who has had a serious adverse reaction to a drug containing the same component as the investigational drug or has a history of allergy
17. Subject who has had a cough, dyspnea, chills, muscle pain, headache, sore throat, loss of smell or taste and an acute fever in which the body temperature exceeds 37.5°C within 72 hours prior to administration of the clinical trial drug
18. Subject who has been diagnosed with COVID-19 and/or have been confirmed or treated for COVID-19 infection as a result of laboratory tests
19. Subject with a history of previous MERS-CoV or SARS-CoV infection
20. Subject with a history of hereditary or idiopathic angioneurotic edema
21. Subject with a history of organ or bone marrow transplantation

    [Relating to contraindicated drugs]
22. Subject who has experience in administering an immunosuppressant or immune modifying drug within 6 months prior to administration of an investigational drug
23. Patients with hemophilia who are at risk of serious bleeding when injected intramuscularly or are taking anticoagulants.
24. Subject who has received immunoglobulin or blood-derived products within 3 months prior to administration of the investigational drug or are expected to administer it during the clinical trial period
25. Subject who participated in other clinical trials similar to the investigational drug before the screening visit (Visit 1)
26. Subject with a history of MERS-CoV or SARS-CoV vaccination
27. Subject who haa received or plan to administer the vaccine within 4 weeks before/after administration of this investigational drug
28. Subject with a history of platelet-related disease or hemorrhagic disease, a history of severe bleeding or bruising after intramuscular injection or venipuncture or a person taking anticoagulants
29. If there is a history of dependent administration of psychotropic drugs or narcotic analgesics within 6 months prior to administration of the investigational drug or in case of a mental illness or social condition in which it is difficult to comply with the clinical trial procedure according to the judgment of the investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events(Immediated AEs) | 30 minutes after each administration
  Incidence rate of immediate adverse events (Immediated AEs)
Adverse event(solicited local / systemic AEs) | 7 days after each administration
  Incidence rate of expected local and systemic adverse events (solicited local / systemic AEs)
Adverse event(unsolicited AEs) | 28 days after each administration
  Incidence rate of unexpected adverse events (unsolicited AEs)
Adverse event(SAEs / serious ADRs) | 28 days after each administration
  Incidence rate of serious adverse events and adverse drug reactions (SAEs / serious ADRs)
Adverse event(AESI) | 394 days from 0 day
  Incidence rate of adverse events of special interest (AESI)

SECONDARY OUTCOMES:
Immunogenicity of QTP104 vaccine as measured by IgG ELISA | Day 0, 29, 57, 180, 394
  Geometric mean titer (GMT) of SARS-CoV-2 Spike (S) protein IgG measured by ELISA at multiple time points after QTP104 administration compared to baseline.
Proportion of subjects for seroconversion of IgG antibodies titer of QTP104 | Day 0, 29, 57, 180, 394
  Proportion of subjects with a ≥4-fold increase in IgG antibody titer to SARS-CoV-2 by ELISA at multiple time points after QTP104 administration compared to baseline.
Immunogenicity of QTP104 vaccine as measured by neutralizing antibodies | Day 0, 29, 57, 180, 394
  Geometric mean titer of neutralizing antibody measured by FRNT using Wild-Type Virus at multiple time points after QTP104 administration compared to baseline

OTHER OUTCOMES:
To analyze the ratio of Th1/Th2 by measuring Th1- and Th2-type cytokines through ICS assay | Day 0, 29, 57, 180, 394
  To analyze the ratio of Th1/Th2 by measuring Th1- and Th2-type cytokines through ICS assay at 4weeks after 1st administration of QTP104 and 4weeks, 5months and 12months after 2nd administration of QTP104
To analyze the cellular immune responses including number of antigen-specific IFN-γ secreting T cells (IFN-γ ELISPOT Assay) | Day 0, 29, 57, 180, 394
  To analyze the cellular immune responses including number of antigen-specific IFN-γ secreting T cells (IFN-γ ELISPOT Assay) at 4weeks after 1st administration of QTP 104 and 4weeks, 5months and 12months after 2nd administration of QTP104

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hwa Choi, Study Director — Quratis Inc.; Joon-Sup Yeom, MD/PhD, Principal Investigator — Infectious Disease, Severance Hospital, Yonsei University College of Medicine; Young Goo Song, MD/PhD, Principal Investigator — Infectious Diseases, Gangnam Severance Hospital, Yonsei University College of Medicine
Locations (2):
- South Korea (2):
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul

REFERENCES:
- See also: korea — http://www.mfds.go.kr